CLINICAL TRIAL: NCT04944758
Title: A Feasibility Study of Adherence to Light Therapy for Maintenance Treatment of Major Depressive Disorder
Brief Title: Feasibility of Adherence to Light Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: We received a grant for an expanded feasibility trial that superseded this one.
Sponsor: University of British Columbia (Other)
Collaborators: Michael Smith Foundation for Health Research (Other)
Responsible Party: Principal Investigator, Raymond Lam, Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V2.0_May-17-2021
Record Dates: First submitted 2021-06-14; First posted 2021-06-30 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Major Depression in Remission
Keywords: major depressive disorder; light therapy; relapse prevention; adherence
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: Open-label feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Light therapy (Other): Daily exposure on weekdays to a standard light device (e.g., fluorescent light box such as the Carex Day-Light Classic, emitting 4000 Kelvin white light rated at 10,000 lux at 14 inches from screen to cornea, with an ultraviolet filter) for 30 minutes as soon as possible after awakening, preferably between 7:00-8:00 am. Participants will also taper and discontinue their antidepressant medication.
  Interventions: Device: Light therapy

INTERVENTIONS:
Device: Light therapy — Light therapy

SUMMARY:
In this feasibility study, we propose an important question: What factors will affect participant adherence to the daily use of light therapy for maintenance treatment of depression? To answer this question, we will conduct a pilot study of open-label treatment with light therapy in a small sample (n=10) of participants meeting eligibility criteria to determine what factors will challenge or enhance adherence to a standard light therapy protocol.

DETAILED DESCRIPTION:
Guidelines recommend at least 6-9 months of maintenance treatment to prevent relapse once patients with major depressive disorder (MDD) are in symptom remission with antidepressant treatment. However, many patients decide to discontinue antidepressants because of side effects or personal preference for a non-pharmacological treatment. Hence, a priority question for patients is whether non-pharmacological treatments can be substituted for antidepressants for maintenance treatment.

Light therapy is a safe, evidence-based, non-pharmacological treatment for MDD and seasonal affective disorder (SAD) with fewer side effects than antidepressants. The safety and efficacy of light therapy suggest that it would also be effective for maintenance treatment and relapse prevention, but there are no studies addressing this question.

Before conducting a randomized controlled trial, we want to determine whether light therapy is feasible for patients in remission with antidepressants and whether patients will adhere to standard light therapy protocols. In this feasibility study, we will enroll patients with MDD in remission who wish to discontinue their antidepressant and substitute open-label light therapy to examine adherence outcomes.

ELIGIBILITY:
Inclusion Criteria:

* [1] Outpatients 19 to 65 years of age;
* [2] Diagnostic and Statistical Manual (DSM)-5 criteria for major depressive disorder (MDD) past or recurrent episode as determined by the Mini International Neuropsychiatric Interview;
* [3] taking an antidepressant for no more than six months;
* [4] participant desire to discontinue antidepressant treatment because of adverse effects or other reasons;
* [5] total score ≤10 on the clinician-rated Montgomery-Asberg Depression Rating Scale [MADRS];
* [6] Willing and able to complete self-report and online assessments including sufficient fluency in English.

Exclusion Criteria:

* [1] Any psychiatric diagnosis other than MDD that is considered the primary diagnosis, including Bipolar I or Bipolar-II (lifetime);
* [2] MDD with psychotic features (lifetime);
* [3] significant personality disorder diagnosis [e.g., borderline, antisocial];
* [4] High suicidal risk, defined by clinician judgment;
* [5] History of drug or alcohol abuse, with a severity of at least moderate or severe within 6 months before screening;
* [6] Significant neurological disorders, head trauma, or other unstable medical conditions;
* [7] regular use of psychotropic medication other than an antidepressant or benzodiazepines (e.g., antipsychotics, mood stabilizers);
* [8] history of severe withdrawal effects with antidepressant discontinuation;
* [9] retinal disease or other eye condition preventing use of bright light therapy;
* [10] use of photosensitizing medication within 1 week of baseline visit.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-04-21 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond W Lam, MD, Principal Investigator — University of British Columbia
Locations (1):
- UBC Mood Disorders Centre, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Light Therapy
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Light Therapy
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 1

OUTCOME MEASURES:

1. Primary Outcome: Adherence Rate
Description: Rate of adherence (>75% of total daily sessions) to light therapy
Time Frame: 6 weeks
Measure: Number; unit: participants
Arm/Group | Light Therapy
Number analyzed (Participants) | 1
participants | 1

2. Secondary Outcome: Relapse Rate
Description: Relapse as defined.
Time Frame: 6 weeks
Population: This is a defined event, "relapse", which is based on several criteria, only one of which is the MADRS scale; however this scale does NOT represent part of the outcome and so is not reported here..
Measure: Count of Participants; unit: Participants
Arm/Group | Light Therapy
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Change in Clinician-rated Depressive Symptoms
Description: Changes in MADRS scores from baseline to 6 weeks (or at relapse or early withdrawal) on the Montgomery-Asberg Depression Rating Scale. MADRS scores range from 0 to 60, with higher scores indicating greater severity of depression (worse outcome).
Time Frame: 6 weeks
Measure: Number; unit: score on a scale
Arm/Group | Light Therapy
Number analyzed (Participants) | 1
score on a scale | 22

4. Secondary Outcome: Change in Patient-rated Depressive Symptoms
Description: Changes in scores from baseline to 6 weeks (or at relapse or early withdrawal) on the Quick Inventory of Depressive Symptomatology, Self-Rated scale (QIDS-SR). The QIDS-SR scores range from 0 to 27, with higher scores indicating greater severity of depression (worse outcome).
Time Frame: 6 weeks
Measure: Number; unit: score on a scale
Arm/Group | Light Therapy
Number analyzed (Participants) | 1
score on a scale | 14

5. Secondary Outcome: Discontinuation Symptoms
Description: Scores on a discontinuation effects scale developed for this study, Antidepressant Discontinuation Symptoms Scale (ADSS). Scores range from 0 to 117, with higher scores indicating more severe discontinuation symptoms (worse outcome).
Time Frame: 4 weeks
Measure: Number; unit: score on a scale
Arm/Group | Light Therapy
Number analyzed (Participants) | 1
score on a scale | 5

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Light Therapy
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Light Therapy (N=1)
Nausea (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Eye strain (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT04944758/Prot_SAP_000.pdf